CLINICAL TRIAL: NCT00501449
Title: Psychosocial Aspects of Multiple Endocrine Neoplasia (MEN) Syndromes
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0783
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Multiple Endocrine Neoplasia
Keywords: Multiple Endocrine Neoplasia; Questionnaire; Psychosocial; Surveillance Behaviors; MEN Syndromes
MeSH Terms: conditions — Multiple Endocrine Neoplasia; Multiple Endocrine Neoplasia Type 1 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Endocrine Neoplasia (MEN): Patients with multiple endocrine neoplasia (MEN).
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Mailed packets including cover letter describing purpose of study, study questionnaire, and return envelope.
  Other Names: Survey

SUMMARY:
The specific aims of the study include:

1. Profile the demographic, health-related, psychosocial and behavioral characteristics of adults with MEN1 or MEN2.
2. Evaluate MEN-specific distress as well as adherence to surveillance regimens among adults with MEN1 or MEN2, and identify associated with those outcomes.

DETAILED DESCRIPTION:
The proposed cross-sectional study is intended to obtain information regarding current surveillance behaviors and other psychosocial outcomes among persons affected by the multiple endocrine neoplasia (MEN) 1 or MEN2, which are inherited conditions.

Study participants will include patients who have been seen previously at MDACC for evaluation of MEN1 or MEN2. Because this is the first time investigators are contacting these patients to invite them to participate in psychosocial research, the proposed study also will help determine the feasibility of conducting similar studies in the future.

Investigators anticipate that data gathered from this study will enhance existing knowledge about the psychological and behavioral aspects of the MEN syndromes, and will inform future research efforts directed toward this understudied population.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 years or older, with a clinical or genetic diagnosis of MEN1 or MEN2
2. Spouse, Significant Other, or Family Member who is at least 18 years of age and who is related to an individual who is a patient at MDACC and who has been diagnosed with MEN1.
3. Ability to read and write English

Exclusion Criteria:

1) Inability to be contacted via mail (i.e., no contact information on record, incorrect address)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of MEN1 or MEN2.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Profile the demographic, health-related, psychosocial and behavioral characteristics of adults with MEN1 or MEN2. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org